CLINICAL TRIAL: NCT04891419
Title: A Multicenter, Evaluator-blinded, Randomized, No-treatment Controlled Study to Evaluate the Safety and Effectiveness of JUVÉDERM® VOLUMA® With Lidocaine for Correction of Temple Hollowing in Chinese Population
Brief Title: JUVÉDERM® VOLUMA® With Lidocaine for Correction of Temple Hollowing in Chinese Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1878-701-008
Record Dates: First submitted 2021-05-14; First posted 2021-05-18 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Temple Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- JUVÉDERM® VOLUMA® with Lidocaine (Experimental): Participants will be treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel in temple. Participants are eligible for touch up treatment
  Interventions: Device: JUVÉDERM® VOLUMA® with Lidocaine
- Control- No treatment (No Intervention): No treatment is administered. Optional treatment at month 6.

INTERVENTIONS:
Device: JUVÉDERM® VOLUMA® with Lidocaine — JUVÉDERM® VOLUMA® with Lidocaine injectable gel
  Arms: JUVÉDERM® VOLUMA® with Lidocaine

SUMMARY:
The objectives of this study are to evaluate the safety and effectiveness of JUVÉDERM® VOLUMA® with Lidocaine injectable gel in adult Chinese population seeking correction of temple hollowing.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 or over, at the time of signing the ICF
* Participants seeking improvement of temple hollowing
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol
* Written informed consent from the participant has been obtained prior to any study-related procedures
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable
* Is able to complete effectiveness self-assessments without the use of glasses (contact lens use is acceptable if they will be used for all participant self-assessments)

Exclusion Criteria:

* Temple hollowing due to trauma, congenital malformations, or lipodystrophy, either congenital or acquired
* Has experienced trauma to the temple area within 6 months before enrollment or has residual deficiencies, deformities, or scarring
* Temporal arteritis or history of temporal arteritis
* Temporomandibular joint dysfunction or any other jaw issues
* Recurrent temporal headaches such as temporal tendinitis migraine
* Active or recurrent inflammation or infection in either eye
* Tendency to develop hypertrophic scarring
* Active autoimmune disease
* History of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), HA products, or Streptococcal protein
* Current cutaneous or mucosal inflammatory or infectious processes (e.g. acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion, above the subnasal
* Prior facial reconstructive surgeries, facelift, or browlift as well as surgeries on the temple area (eg, biopsy)
* Fat injection or permanent facial implants anywhere in the face
* Semipermanent soft-tissue filler treatment in the temple or mid-face within 36 months before enrollment
* Temporary dermal filler injections above the subnasale within 12 months before enrollment
* Mesotherapy or cosmetic facial procedures above the subnasale within 6 months before enrollment (examples of mesotherapy or cosmetic facial procedures are laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures.
* Injections in the nasolabial fold are acceptable only if done at least 3 months prior to enrollment
* Botulinum toxin treatment above the subnasale within 6 months before enrollment
* Has braces or other orthodontics
* Not eligible for this study if participants have begun using any new over the counter or prescription oral or tropical, anti-wrinkle products above the subnasale within 30 days before enrollment. Participants who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study
* Is on a regimen of anti-coagulation therapy (eg, warfarin, clopidogrel)
* Has tattoos, piercings, facial hair, or scars above and including the subnasale that would interfere with visual assessment of the temple
* Females who are pregnant, nursing, or planning a pregnancy
* Plans a significant weight change (more than 10% of body weight) during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN, INC., Study Director — Allergan
Locations (8):
- China (8):
  - China-Japan Friendship Hospital /ID# 241680, Beijing, Beijing Municipality
  - Beijing Hospital /ID# 233582, Beijing, Beijing Municipality
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 233602, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 233607, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 233604, Nanjing, Jiangsu
  - Shanghai Ninth People's Hospital,Shanghai Jiaotong University School of Medicine /ID# 233571, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital /ID# 233568, Shanghai, Shanghai Municipality
  - Peking University International Hospital /ID# 242166, Beijing

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 168 participants were enrolled and randomized (2:1 ratio) to a 12-month treatment group or a 6-month no-treatment group. Participants who completed the no-treatment group had the option to move to a post-control 6-month treatment group. A total of 112 participants were randomized to the 12-month treatment (JUVÉDERM® VOLUMA® with Lidocaine) group and 56 participants were initially randomized to the no-treatment control group.
Groups:
- JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12): Participants will be treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel in temple. Participants are eligible for touch-up treatment.
- Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12): No treatment is administered during the Control No-Treatment period (Months 1 to 6). Only those participants that opt to go on to the Control Treatment period will be treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel in temple.
Period: Overall Study
Arm/Group | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12) | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12)
Started | 112 | 56
Completed the Control Period (Month 1 to 6) | 107 | 56 (Of the 56 completers, 53 moved on to the 6-month post-control treatment.)
Completed the Post Control Period (Months 7 to 12) | 107 | 53
Completed | 107 | 53
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12) | Total
Number analyzed (Participants) | 56 | 112 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (8.16) | 37.3 (9.22) | 36.5 (8.93)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 43 | 75 | 118
  40 - 65 years | 13 | 35 | 48
  > 65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 103 | 156
  Male | 3 | 9 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 56 | 112 | 168
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Allergan Temple Hollowing Scale [Count of Participants; unit: Participants] — Temple with worse baseline score will be used to represent the participant.
  Participants
    Minimal | 22 | 42 | 64
    Moderate | 29 | 62 | 91
    Severe | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug and no more than 30 days after the last dose of the study drug.
Time Frame: Up to 14 Months
Population: Control Period - Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12)
Number analyzed (Participants) | 56 | 112
Participants
  Any TEAE | 23 | 59
  TESAE | 1 | 2

2. Primary Outcome: Participants With at Least a 1-Point Improvement (Decrease) in Temple as Assessed by the Evaluating Investigator (EI) Using the Allergan Temple Hollowing Scale (ATHS)
Description: The Evaluating Investigator will assess the participant's temple hollowing using the ATHS 5-point scale where: 0=convex, rounded temple to 4=severe, deeply recessed, sunken appearance. A 1-point decrease from Baseline indicates improvement.
Time Frame: Change from Baseline to Month 6
Population: Control Period - Observed Primary Endpoint Population
  N = Participants with analysis values at both baseline and Month 6 Visit.
Measure: Number; unit: participants
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12)
Number analyzed (Participants) | 56 | 101
participants | 0 | 92
Statistical Analysis 1: Comparison: Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) vs JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12); Test type: Superiority; p < .0001, Fisher Exact — P-value is based on the Fisher's Exact Test; Rate Difference = 91.1, 95% CI 2-sided [83.7 to 95.9] — 95% exact unconditional confidence interval for between-group difference in responder rate

3. Secondary Outcome: Change From Baseline on Rasch Transformed Score of FACE-Q Satisfaction With Temples Questionnaire at Month 6
Description: Participant-assessed satisfaction using the 12-item FACE-Q Satisfaction with Temples Questionnaire was measured on a 4-point scale where 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, and 4=very satisfied. The responses to the items were converted to a 100-point Rasch transformed score ranging from 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: Change from Baseline to Month 6
Population: Control Period - Modified Intent-to-Treat Population
  N = Participants with analysis values at both baseline and the specified analysis visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12)
Number analyzed (Participants) | 56 | 101
units on a scale | 0.1 (13.97) | 50.7 (26.06)
Statistical Analysis 1: Comparison: Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) vs JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12); Test type: Superiority; p < .0001, Mixed Models Analysis — P-value estimated using mixed effects model; Control Difference = 54.5, 95% CI 2-sided [49.2 to 59.9], Standard Error of Mean 2.69 — 95% CI estimated using mixed effects model

4. Secondary Outcome: Change From Baseline on Rasch Transformed Score of FACE-Q Satisfaction With Facial Appearance Questionnaire at Month 6
Description: Participant-assessed satisfaction using the 10-item FACE-Q Satisfaction with Facial Appearance Questionnaire was measured on a 4-point scale where 1=very dissatisfied, 2=somewhat dissatisfied, 3=somewhat satisfied, and 4=very satisfied. The responses to the items were converted to a 100-point Rasch transformed score ranging from 0 (worst) to 100 (best). Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: Change from baseline to Month 6
Population: Control Period - Modified Intent-to-Treat Population
  Participants with analysis values at both baseline and the specified analysis visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12)
Number analyzed (Participants) | 56 | 101
units on a scale | -4.1 (13.32) | 36.2 (26.89)
Statistical Analysis 1: Comparison: Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) vs JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12); Test type: Superiority; p < .0001, Mixed Models Analysis — 95% CI and p-value estimated using mixed effects model; Control Difference = 42.8, 95% CI 2-sided [37.6 to 48.0], Standard Error of Mean 2.63

5. Secondary Outcome: Participants "Improved" or "Much Improved" as Self-assessed by Participant Using the Global Aesthetic Improvement Scale (GAIS)
Description: Participant will assess temple area using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and-2=much worse.
Time Frame: Month 6
Population: Control Period - Modified Intent-to-Treat Population
  Participants with analysis values at both baseline and the specified visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12)
Number analyzed (Participants) | 56 | 101
Participants | 0 | 94
Statistical Analysis 1: Comparison: Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) vs JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12); Test type: Superiority; p < .0001, Fisher Exact — P-value is based on Fisher's Exact Test; Rate Difference = 93.1, 95% CI 2-sided [86.1 to 97.2] — 95% exact unconditional confidence interval for between-group difference in responder rate

6. Secondary Outcome: Participants "Improved" or "Much Improved" as Assessed by the Evaluating Investigator Using the Global Aesthetic Improvement Scale (GAIS)
Description: The Evaluating Investigator will assess the participant's temple area using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and-2=much worse.
Time Frame: Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) | JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12)
Number analyzed (Participants) | 56 | 101
Participants | 0 | 93
Statistical Analysis 1: Comparison: Control No-Treatment (Months 1 to 6) to JUVÉDERM® VOLUMA® With Lidocaine Treatment (Months 7 to 12) vs JUVÉDERM® VOLUMA® With Lidocaine (Treatment Months 1 - 12); Test type: Superiority; p < .0001, Fisher Exact — P-value is based on Fisher's Exact Test; Rate Difference = 92.1, 95% CI 2-sided [84.9 to 96.5] — 95% exact unconditional confidence interval for between-group difference in responder rate

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 6.4, 12.8 and 6.9 months for No Treatment (Control Period), JUVÉDERM® VOLUMA® with Lidocaine (Treatment Period), and JUVÉDERM® VOLUMA® with Lidocaine (Post-Control Treatment Period), respectively.
Groups:
- Control - No Treatment (Months 1 - 6): No treatment is administered. Optional treatment at Month 6.
- JUVÉDERM® VOLUMA® With Lidocaine (Months 1 - 12): Participants will be treated with JUVÉDERM® VOLUMA® with Lidocaine injectable gel in temple. Participants are eligible for touch-up treatment.
- JUVÉDERM® VOLUMA® With Lidocaine - Post Control (Months 7 - 12): Participants will be treated with optional JUVÉDERM® VOLUMA® with Lidocaine injectable gel in temple through study exit date.
Arm/Group | Control - No Treatment (Months 1 - 6) | JUVÉDERM® VOLUMA® With Lidocaine (Months 1 - 12) | JUVÉDERM® VOLUMA® With Lidocaine - Post Control (Months 7 - 12)
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/112 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/56 | 3/112 | 2/53
Other Adverse Events (participants affected / at risk) | 18/56 | 62/112 | 19/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control - No Treatment (Months 1 - 6) (N=56) | JUVÉDERM® VOLUMA® With Lidocaine (Months 1 - 12) (N=112) | JUVÉDERM® VOLUMA® With Lidocaine - Post Control (Months 7 - 12) (N=53)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control - No Treatment (Months 1 - 6) (N=56) | JUVÉDERM® VOLUMA® With Lidocaine (Months 1 - 12) (N=112) | JUVÉDERM® VOLUMA® With Lidocaine - Post Control (Months 7 - 12) (N=53)
INJECTION SITE PAIN (General disorders) | 0 (0) | 11 (34) | 1 (4)
INJECTION SITE SWELLING (General disorders) | 0 (0) | 7 (17) | 1 (2)
COVID-19 (Infections and infestations) | 18 (18) | 47 (47) | 13 (14)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 6 (6) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
TRISMUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8) | 4 (4)
DIZZINESS (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04891419/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT04891419/SAP_001.pdf